CLINICAL TRIAL: NCT00255450
Title: A Double Blind, Placebo Controlled, Crossover Design, Multicenter Study of Intravenous Ferumoxytol Compared With Placebo
Brief Title: A Crossover Safety Study of Ferumoxytol Versus Placebo
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AMAG Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 62745-8
Record Dates: First submitted 2005-11-17; First posted 2005-11-21 (Estimated); Last update posted 2008-11-11 (Estimated); Status verified 2007-10

CONDITIONS: Anemia
Keywords: anemia
MeSH Terms: conditions — Anemia | interventions — Ferrosoferric Oxide

INTERVENTIONS:
Drug: ferumoxytol or placebo

SUMMARY:
This crossover safety study will evaluate the safety of a single dose of ferumoxytol compared to placebo in patients with chronic kidney disease.

DETAILED DESCRIPTION:
This is a double-blind, placebo controlled, crossover design study of the safety of ferumoxytol compared to placebo. Patients are randomized to receive either one 510 mg dose of ferumoxytol or the equivalent volume of normal saline followed by the other test article given one week later.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients > 18 years.
* Have chronic kidney disease per K/DOQI guidelines.
* Baseline hemoglobin of > 9.0 and < 12.5 g/dl

Exclusion Criteria:

* Women who are pregnant or lactating.
* Received another investigational drug or device within 30 days.
* Recent parenteral or oral iron therapy.
* Patients that have other causes of anemia.
* Major surgery within 30 days or anticipated or planned surgery during the study.
* Patients with active infections.
* Recent blood transfusions.
* Patients with known allergies to iron products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750
Dates: Start 2005-01; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Safety evaluated by physical examinations, vital signs, laboratory tests and patient monitoring and evaluation.

CONTACTS AND LOCATIONS:
Locations (39):
- United States (39):
  - Mobile, Alabama
  - Phoenix, Arizona
  - Mountain View, California
  - New Haven, Connecticut
  - Washington D.C., District of Columbia
  - Ocala, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Newnan, Georgia
  - Peoria, Illinois
  - Shreveport, Louisiana
  - Bethesda, Maryland
  - Boston, Massachusetts
  - Detroit, Michigan
  - St Louis, Missouri
  - Broken Bow, Nebraska
  - Lebanon, New Hampshire
  - Flushing, New York
  - New York, New York
  - Orchard Park, New York
  - Raleigh, North Carolina
  - Columbus, Ohio
  - Portland, Oregon
  - Erie, Pennsylvania
  - Lancaster, Pennsylvania
  - Greenville, South Carolina
  - Sumter, South Carolina
  - Chattanooga, Tennessee
  - Knoxville, Tennessee
  - Austin, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Alexandria, Virginia
  - Charlottesville, Virginia
  - Chesapeake, Virginia
  - Norfolk, Virginia
  - Bluefield, West Virginia
  - Appleton, Wisconsin

REFERENCES:
- [Background] Landry R, Jacobs PM, Davis R, Shenouda M, Bolton WK. Pharmacokinetic study of ferumoxytol: a new iron replacement therapy in normal subjects and hemodialysis patients. Am J Nephrol. 2005 Jul-Aug;25(4):400-10. doi: 10.1159/000087212. Epub 2005 Jul 28. PMID 16088081
- [Result] Singh A, Patel T, Hertel J, Bernardo M, Kausz A, Brenner L. Safety of ferumoxytol in patients with anemia and CKD. Am J Kidney Dis. 2008 Nov;52(5):907-15. doi: 10.1053/j.ajkd.2008.08.001. Epub 2008 Sep 27. PMID 18824288
- [Derived] Natale P, Ju A, Strippoli GF, Craig JC, Saglimbene VM, Unruh ML, Stallone G, Jaure A. Interventions for fatigue in people with kidney failure requiring dialysis. Cochrane Database Syst Rev. 2023 Aug 31;8(8):CD013074. doi: 10.1002/14651858.CD013074.pub2. PMID 37651553
- See also: National Kidney Foundation — http://www.kidney.org/index.cfm